CLINICAL TRIAL: NCT06141863
Title: Investigation of Temporomandibular Dysfunction in Patients With Cervical Disc Herniation
Brief Title: Temporomandibular Dysfunction in Patients With Cervical Disc Herniation
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Turgay Altunalan, Assist Professor, Karadeniz Technical University
Other Study IDs: 6135131342/2022-28
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Temporomandibular Joint Dysfunction Syndrome; Intervertebral Disc Displacement; Disability; Neck; Jaw
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Intervertebral Disc Displacement | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: no disability and mild disability
  Interventions: Other: questionnaire
- Group 2: moderate and severe disability
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Neck Disability Index, The Fonseca Anamnestic Index (FAI) and Visual Analogue Scale (VAS)

SUMMARY:
Cervical spine problems are associated with temporomandibular joint (TMJ) and related muscles.The aim of the present study was to investigate temporomandibular joint dysfunction (TMD) and pain in individuals with cervical disc herniation (CDH) according to the level of neck disability.

DETAILED DESCRIPTION:
The study included diagnosed with cervical disc herniation. The participants were divided into two groups based on their The Neck Disability Index (NDI) score: Group 1 with no disability and mild disability and Group 2 with moderate and severe disability. Temporomandibular dysfunction and its severity, intensity of neck and temporomandibular joint pain was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical disc herniation aged between 18 and 65,
* who could read and write in Turkish

Exclusion Criteria:

* Individuals with a history of head and neck surgery, fracture, physiotherapy or medical treatment cervical or temporomandibular joint treatment within the last six months,
* presence of any inflammatory rheumatic diseases, such as ankylosing spondylitis and rheumatoid arthritis, facial paralysis, infection, advanced osteoporosis

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with cervical disc herniation. Patients who were referred to physiotherapy after diagnosis were evaluated in terms of study suitability before starting treatment. We divided the participants into two groups based on their level of neck disability to compare their TMD.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | one day assessment
  Assessment of neck disability
Fonseca Anamnestic Index | one day assessment
  Assessment of temporomandibular dysfunction

SECONDARY OUTCOMES:
Visual Analogue Scale | one day assessment
  Assessment of temporomandibular joint pain and neck pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Turgay Altunalan, Assist Prof, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)